CLINICAL TRIAL: NCT02835391
Title: A Prospective, Multi-Centre, Randomized, Safety and Effectiveness Study of PerClot Compared to Usual Care When Used During Gynaecology Procedures
Brief Title: PerClot Compared to Usual Care in Gynaecology Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CryoLife Europa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCT1501-000-C(01/15)
Record Dates: First submitted 2015-07-31; First posted 2016-07-18 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2016-07

CONDITIONS: Endometriosis; Ovarian Cyst; Menorrhagia; Cancer; Uterine Fibroids
MeSH Terms: conditions — Endometriosis; Ovarian Cysts; Menorrhagia; Neoplasms; Leiomyoma | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PerClot (Active Comparator): PerClot® Polysaccharide Hemostatic System (PerClot) is a medical device composed of absorbable polysaccharide particles (AMPs) and delivery applicators. Investigators will have the option to choose 3g or 5g dependent on the requirements of the patient
  Interventions: Device: PerClot
- Usual Care (Active Comparator): Usual care will consist of any other haemostat the Investigator would normally use in the control of bleeding i.e arista, Floseal, surgical, surgiflo. If the Investigator would not normally use a haemostat to control bleeding then electrocautery or diathermy may be used in this arm
  Interventions: Device: Floseal, Surgicel, Surgiflo, Arista; Procedure: Electrocautery/Diatermy

INTERVENTIONS:
Device: PerClot — Haemostatic device for the control of bleeding from capillary, venous or arteriolar vessels by pressure, ligature or other conventional means is either ineffective or impractical.
  Arms: PerClot
Device: Floseal, Surgicel, Surgiflo, Arista — Haemostatic device for the control of bleeding
  Arms: Usual Care
Procedure: Electrocautery/Diatermy — Procedure for the control of bleeding
  Arms: Usual Care

SUMMARY:
This study is a post market, multi-centre, randomised study evaluating PerClot compared to usual care. PerClot is a CE marked device and is currently used as a haemostat in gynaecological surgery throughout Europe. The purpose of this study is to collect additional post market data on its use in this indication.

DETAILED DESCRIPTION:
This study is a post market, multi-centre, randomised study evaluating PerClot compared to usual care.

All subjects in this randomized study will undergo a laparoscopic or open gynecological procedure such as hysterectomy, cystectomy, myomectomy, endometrial excision or ablation. Subjects will be randomized to receive PerClot or usual care.

This research will utilize a multi-center, prospective, randomized controlled study. The study will be conducted in2 study sites in Europe. An assumed sample of 90 subjects will be enrolled to evaluate the time to haemostasis. The enrollment of subjects to receive treatment will be based upon specific inclusion and exclusion criteria. Subjects will be randomized on a 1:1 basis to receive either PerClot or usual care. Data collected from both arms will be compared.

Usual care will be at the discretion of the surgeon and may include any other haemostat or diathermy/electrocautery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is undergoing gynecological procedure
* Subject is willing and able to comply with the protocol and follow up period
* Subject is willing and able to give written informed consent

Exclusion Criteria:

* • Subject with a history of pelvic or abdominal radiotherapy (within 8 weeks)

  * Subject is pregnant or actively breastfeeding
  * Subject has a ruptured ectopic pregnancy
  * Subject has a medical history of abnormal coagulopathy or bleeding
  * Subject has a sensitivity to starch or starch derived materials
  * Subject has active or potential infection at the surgical site
  * Subject is currently enrolled in another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
achievement of haemostasis (yes/no). | measured up to 10 minutes after application
  visual observation of cessation of bleeding

SECONDARY OUTCOMES:
Absence of re-intervention for post-operative bleeding | within 30 days of initial surgery
  No return to OR for bleeding

OTHER OUTCOMES:
Absence of proven infection | within 30 days of initial surgery
  No positive culture of blood results which indicate infection
Absence of bleeding related adverse events | within 30 days of initial surgery
  No adverse events which are specifically caused by bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Bellvitge Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ponce J, Garcia-Tejedor A, Barahona M, Cappuccio S, Costantini B, Fedele C, Marti-Cardona L, Scambia G. Effectiveness and safety of an absorbable modified polymer starch powder hemostat versus usual care in gynecology procedures: A prospective, multi-center, and randomized study. PLoS One. 2025 Sep 11;20(9):e0331376. doi: 10.1371/journal.pone.0331376. eCollection 2025. PMID 40934160